CLINICAL TRIAL: NCT05319613
Title: Reducing Disparities in Rural HIV Prevention With Telemedicine PrEP and Postal Lab Kits
Brief Title: Reducing Disparities in Rural HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-2514
Record Dates: First submitted 2022-03-11; First posted 2022-04-08 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: HIV Infections; Sexually Transmitted Infections
Keywords: HIV Prevention, Access, Rural Communities
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Convenience sample of baseline community survey participants who elect to enter clinical PrEP care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine Clinical Care (Other): Rural participants who enter PrEP clinical care with University of Colorado HIV Prevention Program will receive care via telemedicine with mailed lab kits and mailed HIV PrEP.
  Interventions: Other: Virtual clinical visits with home lab kits and mailed HIV PrEP

INTERVENTIONS:
Other: Virtual clinical visits with home lab kits and mailed HIV PrEP — Rural participants who enter PrEP care with University of Colorado HIV Prevention Program will receive PrEP services via telemedicine with home lab kits and mailed HIV PrEP

SUMMARY:
HIV and Sexually Transmitted Infection (STI) rates are increasing in rural areas including rural Colorado. Many rural residents find it difficult to access HIV and STI prevention services.

In this study, an online survey on HIV and STI Prevention and best practices to provide access to prevention will be administered to rural residents in three zip 3 zones in rural Colorado. In addition to the baseline survey, study participants who are interested and medically eligible may initiate PrEP services with the University of Colorado HIV Prevention Program and receive PrEP through telemedicine visits, mailed home lab kits, and mailed medication. Persistence in PrEP care, acceptability, and feasibility of telemedicine and home lab kits will be measured.

DETAILED DESCRIPTION:
HIV and Sexually Transmitted Infection (STI) rates are increasing in rural areas including rural Colorado. Many rural residents find it difficult to access HIV and STI prevention services. The goal of this study is to understand the risk for HIV and STIs, views on PrEP, and to determine if access to telemedicine visits and home lab kits increases engagement in PrEP services and persistence in care for at-risk rural populations.

An online survey on HIV and STI Prevention and best practices to provide access to prevention will be administered to rural residents in three zip 3 zones in rural Colorado, comprised of increased proportions of minority residents (Hispanic, Native American, and Black). In addition to the baseline survey, study participants who are interested and medically eligible may initiate PrEP services with the University of Colorado HIV Prevention Program and receive PrEP through telemedicine visits, mailed home lab kits, and mailed medication. Persistence in PrEP care, acceptability, and feasibility of telemedicine and home lab kits will be measured through baseline and follow-up survey questionnaires and clinical chart reviews for those engaged in PrEP care.

ELIGIBILITY:
Inclusion Criteria:

1. Colorado rural or frontier county residents, Adults (age 18+)
2. Access to internet, smart phone or tablet to participate in online surveys
3. Able to complete online surveys in English or Spanish

Exclusion Criteria:

1. Residence in an urban Colorado county
2. HIV positive status
3. No internet, smart phone, or tablet access
4. Unable to complete online surveys in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Persistence in PrEP care | 12 months
  The proportion of study participants persisting in PrEP care at 12 months, stratified by race, ethnicity, zip 3 region, and type of insurance coverage.

SECONDARY OUTCOMES:
Medication adherence | 12 months
  Describe PrEP medication adherence rates at 12 months (as determined by pharmacy refill data) for rural CO PrEP users who utilize Telemedicine PrEP services and postal lab kits.
Feasibility of Telemedicine visits | 12 months
  Describe feasibility of Telemedicine visits as determined by survey response and completion of quarterly visits.
Acceptability of Telemedicine visits | 12 months
  Describe acceptability of Telemedicine visits as determined by survey response and completion of quarterly visits.
Feasibility of postal lab kits | 12 months
  Describe feasibility of postal lab kits, as determined by survey response and completion of quarterly lab monitoring.
Acceptability of postal lab kits | 12 months
  Describe acceptability of postal lab kits, as determined by survey response and completion of quarterly lab monitoring.
HIV seroconversion | 12 months
  Describe rate of HIV seroconversion in cohort at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. De-identified aggregate data will be shared at completion of study.